CLINICAL TRIAL: NCT04644042
Title: The Effect of Arthroscopic Subacromial Decompression in Patients With Subacromial Impingement Syndrome Who Are Non-responders to Non-operative Treatment. A Double-blinded, Randomized, Controlled Trial.
Brief Title: The Effect of Arthroscopic Subacromial Decompression in Patients Who Are Non-responders to Non-operative Treatment.
Acronym: SELECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Adam Witten, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SELECT trial
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glenohumeral arthroscopy and arthroscopic subacromial decompression (Experimental): The intervention group will receive a glenohumeral arthroscopy and ASAD. Participants are discharged with an arm sling and referred to 3 months physiotherapy in a municipally setting. Participants are given a rehabilitation program containing progressive exercises to guide the rehabilitation.
  Interventions: Procedure: Glenohumeral arthroscopy + Arthroscopic Subacromial Decompression
- Glenohumeral arthroscopy and skin incision (Active Comparator): The control group will receive a glenohumeral arthroscopy, but no treatment concerning the subacromial structures. To allow for the best possible blinding, a 7-10 mm incision, mimicking the one used for ASAD, is performed on the lateral side of the arm 2-3 distal to the acromion. Participants are discharged with an arm sling and referred to 3 months physiotherapy in a municipally setting. Participants are given a rehabilitation program containing progressive exercises to guide the rehabilitation.
  Interventions: Procedure: Glenohumeral arthroscopy + lateral skin incision

INTERVENTIONS:
Procedure: Glenohumeral arthroscopy + Arthroscopic Subacromial Decompression — In addition to the glenohumeral athroscopy a lateral portal will be used to access the subacromial space. The subacromial space will be decompressed with removal of inflamed bursal tissue and acromioclavicular osteophytes, release of the coracoacromial ligament, and, if deemed necessary by the surgeon, acromioplasty performed ad modum Caspari.
  Arms: Glenohumeral arthroscopy and arthroscopic subacromial decompression
Procedure: Glenohumeral arthroscopy + lateral skin incision — Glenohumeral arthroscopy is performed as a standard investigational procedure. The patient is put under general anesthesia and positioned in the 'beach chair position'. An anteriorsuperior portal and a posterior mid-glenoid portal are used as entry to the joint. The following structures are investigated as a minimum: the articular surface of the humeral head and the glenoid, labrum, the long biceps tendon and its attachment at the superior labrum, the undersurface of the supraspinatus and the infraspinatus tendon, the subscapularis tendon and the glenohumeral ligaments. To allow for the best possible blinding a skin incision (mimicking the one used for arthroscopic subacromial decompression) is performed on the lateral side of the shoulder of the participants in the control group. The obturator is introduced in the subcutaneous tissue and a slight circular release is performed. The deltoid fascia is not perforated and the subacromial space is not entered.
  Arms: Glenohumeral arthroscopy and skin incision

SUMMARY:
To investigate if glenohumeral arthroscopy and arthroscopic subacromial decompression is more effective than glenohumeral arthroscopy alone in improving patient-reported outcome at 12 months in patients with subacromial impingement syndrome (SIS) who are non-responders to non-operative treatment.

DETAILED DESCRIPTION:
The trial is designed as a patient and assessor-blinded, randomized, controlled trial with two parallel groups. Participants are randomized 1:1 to either ASAD and glenohumeral arthroscopy (intervention group) or glenohumeral arthroscopy alone (control group). The two groups are subscribed identical postoperative rehabilitation consisting of 3 months physiotherapy in a municipally setting. The primary endpoint is the Shoulder Pain and Disability Index (SPADI) 12 months after surgical intervention. The study will adhere to the CONSORT guidelines.

All participants will be recruited consecutively from the outpatient clinic, Arthroscopic Center, Copenhagen University Hospital, Hvidovre. Consultant orthopedic surgeons will conduct the initial eligibility screening as part of their consultation. Eligible participants will be provided with thorough verbal and written information about the trial and their right to withdraw at any time. Patients given their written, informed consent to participate in the trial, will receive scheduled appointments for the baseline examination.

ELIGIBILITY:
Inclusion Criteria:

* SIS diagnosis (Consultant's clinical diagnosis of SIS + at least 3 out of 5 positive tests from the following: Hawkin's, Neer's, Jobe's, Painful arc and external rotation resistance test)
* Positive subacromial injection test
* Insidious onset of shoulder pain
* Considered a surgical candidate by an orthopedic shoulder specialist.
* Symptoms for at least 6 months
* Completion of at least 3 months supervised shoulder training
* No improvement in symptoms for at least 3 months
* The patient must be expected to be able to attend rehabilitation and post-examinations.

Exclusion Criteria:

* Terminal illness or severe medical illness (ASA score higher than or equal to 4), systemic musculoskeletal disease, inflammatory joint disease (e.g. rheumatoid arthritis), symptomatic cervical spine pathology or thoracic outlet syndrome.
* Full-thickness rotator cuff tear, calcified tendonitis, labral tear, frozen shoulder, biceps tendon pathology, acromioclavicular osteoarthrosis, glenohumeral osteoarthrosis or other concomitant shoulder pathology.
* Previous surgery or radiotherapy on the affected shoulder.
* Pregnancy
* Ongoing workers compensation case or job rehabilitation process

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | 12 months after surgical intervention.
  The primary outcome is SPADI 12 months after surgical intervention.

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | 24 months
  SPADI is registered as a secondary outcome 3, 6 and 24 months after surgical intervention.
Oxford Shoulder Score | 24 months
  Oxford Shoulder Score is registered 3, 6, 12 and 24 months after surgical intervention.
Patient Satisfaction | 12 months
  Patient satisfaction will be assessed using three questions:
  1. "How are the problems related to your shoulder now, compared with before surgery?" (response options: no problems at all, much better, slightly better, no change, slightly worse, much worse)
  2. "Overall, how pleased have you been with the result of your surgery so far?" (response options: very pleased, fairly pleased, not very pleased, very disappointed)
  3. "If you could go back in time, would you still choose to have the shoulder operation?" (response options: yes, no, not sure).
Active Shoulder Abduction Range Of Motion (AROM) | 12 months
  Active Shoulder Abduction Range Of Motion is registered at 3 and 12 months after surgical intervention.
Pain during Active Shoulder Abduction Range Of Motion (NPRS-AROM) | 12 months
  Pain during active shoulder abduction range of motion is evaluated using the numeric pain rating scale (NPRS) at 3 and 12 months after surgical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kristoffer Barfod, MD, Study Director — Sports Orthopedic Research Center - Copenhagen (SORC-C), Hvidovre Hospital
Locations (1):
- Hvidovre Univeristy Hospital, Hvidovre, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No